CLINICAL TRIAL: NCT04458922
Title: A Phase 2 Study of Anti-PD-L1 Antibody (Atezolizumab) in Chondrosarcoma and Clear Cell Sarcoma
Brief Title: Testing Atezolizumab in People 2-17 Years Old With Clear Cell Sarcoma or Advanced Chondrosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-04634; NCI-2020-04634 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 000081; 20-C-XXXX; 10398 (Other: National Cancer Institute LAO); 10398 (Other: CTEP)
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-06

CONDITIONS: Central Chondrosarcoma, Grade 2; Central Chondrosarcoma, Grade 3; Dedifferentiated Chondrosarcoma; Metastatic Clear Cell Sarcoma of Soft Tissue; Metastatic Primary Central Chondrosarcoma; Unresectable Primary Central Chondrosarcoma
MeSH Terms: conditions — Lymphoma, Follicular; Sarcoma, Clear Cell | interventions — atezolizumab; Biopsy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atezolizumab) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on ay 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scans and undergo biopsy and collection of blood samples on study.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biopsy Procedure — Correlative studies
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography

SUMMARY:
This phase II trial studies how well atezolizumab works in treating patients with chondrosarcoma or clear cell sarcoma that is newly diagnosed, cannot be removed by surgery (unresectable), or has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the objective response rates (ORR) using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 of atezolizumab in adult (>= 18 years) patients with clear cell sarcoma (CCS) and chondrosarcoma (CS).

SECONDARY OBJECTIVES:

I. Determine duration of response (DOR) using RECIST v 1.1 and/or change in clinical symptoms (time frame: baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination).

II. Measure progression-free survival (PFS) time (time frame: baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination).

III. Assess the number of activated CD8+ T cells infiltrating the tumor before and after atezolizumab treatment, and correlate treatment-induced changes with clinical response.

EXPLORATORY OBJECTIVES:

I. Compare RECIST v 1.1 versus (vs) immune RECIST (iRECIST) in patients with CCS and CS on atezolizumab.

II. Examine changes in PD-1/PD-L1 expression in the tumor microenvironment before and after atezolizumab treatment, and correlate treatment-induced changes with clinical response.

III. Evaluate potential associations between atezolizumab activity and tumor genomic alterations.

OUTLINE:

Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scans and undergo biopsy and collection of blood samples on study.

After completion of study treatment, patients are followed up to 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented EWSR1/ATF1 or EWSR1/CREB1 translocation or histologically confirmed clear cell sarcoma, documented grade 2 or 3 conventional chondrosarcoma, or documented dedifferentiated chondrosarcoma. The disease must not be curable by surgery
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients with newly diagnosed, unresectable, metastatic and measurable clear cell sarcoma, EWSR1/ATF1 or EWSR1/CREB1 translocation, grade 2 or 3 conventional chondrosarcoma, or dedifferentiated chondrosarcoma will also be eligible if they show clinical evidence of disease progression (including history and increasing physical symptoms). On-study documentation will include a physician's rationale that supports evidence of clinical disease progression (i.e., increasing tumor pain)
* Age >= 2 years at the National Cancer Institute (NCI) Clinical Center (>= 12 years at other participating sites)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky or Lansky >= 70%)
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8 g/dL
* Total bilirubin =< institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN (AST and/or ALT =< 5 x ULN for patients with liver involvement)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN for patients with documented liver involvement or bone metastases)
* Creatinine:

  * For adult patients (>= 18 years of age): >= 30 mL/min/1.73 m^2 by Cockcroft-Gault
  * For pediatric patients (< 18 years of age), a serum creatinine based on age and gender as follows:

    * Age: 2 to < 6 years; Maximum serum creatinine (mg/dL): 0.8 (male) 0.8 (female)
    * Age: 6 to < 10 years; Maximum serum creatinine (mg/dL): 1 (male) 1 (female)
    * Age: 10 to < 13 years; Maximum serum creatinine (mg/dL): 1.2 (male) 1.2 (female)
    * Age: 13 to < 16 years; Maximum serum creatinine (mg/dL): 1.5 (male) 1.4 (female)
    * Age: 16 to < 18 years; Maximum serum creatinine (mg/dL): 1.7 (male) 1.4 (female)
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for >= 1 month after treatment of the brain metastases
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS-specific treatment is not required and is unlikely to be required during the first 2 cycles of therapy
* Patients with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Willingness to provide biopsy samples for research purposes (patients >= 18 years of age only)
* Administration of atezolizumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality. Female patients of child-bearing potential and male patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document or a parent/guardian able to do the same

Exclusion Criteria:

* Any prior therapy must have been completed >= 4 weeks or, if known, >= 5 half-lives of the prior agent (whichever is shorter) prior to enrollment on protocol (minimum of 1 week between prior therapy and study enrollment), and the participant must have recovered to eligibility levels from prior toxicity. Patients should be at least 6 weeks out from nitrosoureas and mitomycin C. Prior definitive radiation should have been completed >= 4 weeks or palliative radiation should have been completed >= 2 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels (patients on study may be eligible for palliative radiotherapy to non-targeted lesions after 2 cycles of therapy at the principal investigator [PI's] discretion). Patients who have had prior monoclonal antibody therapy must have completed that therapy >= 6 weeks (or 3 half-lives of the antibody, whichever is shorter) prior to enrollment on protocol (minimum of 1 week between prior therapy and study enrollment). A patient who has received a cumulative dose of > 350 mg/m^2 of anthracycline (regardless of cardioprotectant) may only be enrolled if their ejection fraction measured by an echocardiogram is within normal institutional limits
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents

  * Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met:

    * Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose
    * No history of severe immune-related adverse effects from anti-CTLA-4 (NCI Common Terminology Criteria for Adverse Events [CTCAE] grade 3 and 4)
* Treatment with any other investigational agent within 4 weeks (or within five half lives of the investigational product, whichever is shorter) prior to cycle 1, day 1 (minimum of 1 week between prior therapy and study enrollment). Patients must be >= 2 weeks since any investigational agent administered as part of a phase 0 study (also referred to as an "early phase I study" or "pre-phase I study" where a sub-therapeutic dose of drug is administered) at the coordinating center PI's discretion, and should have recovered to eligibility levels from any toxicities
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon-alpha or interleukin-2 [aldesleukin]) within 6 weeks prior to cycle 1, day 1
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone [ > 10 mg/day], cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1.

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids and systemic mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia. Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies (i.e., antibodies with generic names ending in "ximab" or "zumab", respectively) or fusion proteins
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because atezolizumab is an investigational agent with the unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atezolizumab, breastfeeding should be discontinued if the mother is treated with atezolizumab
* Patients with a history of human immunodeficiency virus (HIV)-positive on antiretroviral therapy are eligible with an undetectable viral load. For those patients, an HIV viral load test must be completed within 28 days prior to enrollment
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease.

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis.

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with autoimmune hyperthyroid disease not requiring immunosuppressive treatment may be eligible
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to cycle 1, day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2025-12-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: A P Chen, Principal Investigator — National Cancer Institute LAO
Locations (15):
- United States (14):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS): Participants with clear cell sarcoma receive atezolizumab intravenous (IV) over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo computed tomography (CT) scans and undergo biopsy and collection of blood samples on study.
- Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3): Participants with conventional chondrosarcoma, grade 2 or 3, receive atezolizumab intravenous (IV) over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo computed tomography (CT) scans and undergo biopsy and collection of blood samples on study.
- Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS): Participants with dedifferentiated chondrosarcoma receive atezolizumab intravenous (IV) over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo computed tomography (CT) scans and undergo biopsy and collection of blood samples on study.
Period: Overall Study
Arm/Group | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS)
Started | 9 | 9 | 9
Completed | 0 | 0 | 1
Not Completed | 9 | 9 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Protocol -specified withdrawal criterion met | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Started new study | 0 | 0 | 1
Not completed — Progressive disease | 6 | 8 | 2
Not completed — Death | 1 | 0 | 2
Not completed — Participant started chemotherapy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS) | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 5 | 21
  >=65 years | 0 | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.11 (7.9) | 52.89 (11.4) | 64.89 (9.57) | 51.63 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 3 | 10
  Male | 4 | 7 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 5 | 7 | 9 | 21
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 6 | 6 | 8 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 0 | 1
  United States | 9 | 8 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates (ORR)
Description: ORR was measured using the Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1, which involves the following response definitions. Complete Response (CR): disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR): at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Progressive Disease (PD): at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Baseline until confirmation of progressive disease or response (complete or partial) as defined by RECIST v1.1, an average of 4 months.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS)
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 33.33 | 33.33 | 33.33
  Progressive Disease | 55.56 | 66.67 | 44.44
  Unknown (not assessed) | 11.11 | 0 | 22.22

2. Secondary Outcome: Duration of Response (DOR) or Change in Clinical Symptoms
Description: Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Complete Response (CR): disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR): at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progression was measured using the Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 and/or change in clinical symptoms. Progressive Disease (PD): is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination, assessed up to 3 years
Population: The analysis population was to include all participants with an objective response (complete or partial). Because no objective responses were observed, there was no evaluable population and data were not collected.
Arm/Group | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Progression-free Survival (PFS) Time
Description: PFS is the time interval from start of treatment to documented evidence of disease progression, measured by the Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1, or death from any cause, whichever comes first. Progressive Disease (PD): at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS)
Number analyzed (Participants) | 9 | 9 | 9
Months | 2.66 [2.04 to NA] — The reason NA is listed as the upper limit of the confidence interval is that "Given the size and distribution of the sample set, there is not sufficient data to estimate the upper bounds." | 3.22 [2.07 to NA] — The reason NA is listed as the upper limit of the confidence interval is that "Given the size and distribution of the sample set, there is not sufficient data to estimate the upper bounds." | 2.04 [1.22 to NA] — The reason NA is listed as the upper limit of the confidence interval is that "Given the size and distribution of the sample set, there is not sufficient data to estimate the upper bounds."

4. Secondary Outcome: Number of Activated Cluster of Differentiation 8 (CD8+) T Cells Infiltrating the Tumor
Description: Activated CD8+ T cells will be detected by multiplex immunofluorescence assays and will be defined by the expression of T cell receptor (TCR) activation (Zeta chain phosphorylation) or phosphorylated Zap70 (pY493); CD8+ cells present within the tumor section that are positive for these markers will be quantified.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2025-12

5. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 22 days, 8 months and 27 days, and 11 months and 22 days for each Arm/Group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS)
Number analyzed (Participants) | 9 | 9 | 9
Participants | 9 | 8 | 9

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 22 days, 8 months and 27 days, and 11 months and 22 days for each Arm/Group respectively.
Description: The descriptions and grading scales found in the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 were utilized for adverse event (AE) reporting. An adverse event that began in one cycle and resolved in another cycle is considered a single adverse event.
Arm/Group | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS)
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/9 | 2/9
Serious Adverse Events (participants affected / at risk) | 5/9 | 1/9 | 6/9
Other Adverse Events (participants affected / at risk) | 9/9 | 8/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) (N=9) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) (N=9) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS) (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Gluteal muscle myonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, abscess- right thigh (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Right sided facial droop (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Immune system disorders - Other, systemic immune activation (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Erythema of the skin on the right buttock (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Atezolizumab 1200 mg Intravenous (IV) on Day 1, Subgroup 1: Clear Cell Sarcoma (CCS) (N=9) | Arm 1 Atezolizumab 1200 mg IV on Day 1, Subgroup 2: Conventional Chondrosarcoma (CS)(Grade 2 or 3) (N=9) | Arm 1 Atezolizumab 1200 mg Intravenous on Day 1, Subgroup 3: Dedifferentiated Chondrosarcoma (CS) (N=9)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 7 (17) | 1 (1) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 7 (11) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (2) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (16) | 1 (1) | 5 (5)
Edema face (General disorders) | 2 (3) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 1 (1) | 2 (2)
Edema trunk (General disorders) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, macular edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (16) | 6 (7) | 1 (1)
Fever (General disorders) | 5 (7) | 1 (1) | 2 (2)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, appetite increased (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (21) | 1 (1) | 4 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 3 (5) | 3 (4) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (9) | 0 (0) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (3)
Investigations - Other, Chloride Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, Hypoprotenemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, Total Protein Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 3 (5) | 3 (3)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Gluteal muscle myonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Myotonic Jerking (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, right hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (2) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (2)
Pain (General disorders) | 3 (6) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3) | 3 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Periorbital edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 2 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Renal and urinary disorders - Other, Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, Swelling Lt inguinal area (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (10) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Blistering over bone hardware (LLE) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Surgical and medical procedures - Other, pleural catheter (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (3) | 1 (1)
Weight loss (Investigations) | 4 (8) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04458922/Prot_SAP_000.pdf
  • Informed Consent Form: Adult Consent (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04458922/ICF_001.pdf
  • Informed Consent Form: Pediatric Consent (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04458922/ICF_002.pdf